CLINICAL TRIAL: NCT04141345
Title: Influence of Comorbid Chronic Lung Disease on Heart Failure Long-Term Outcomes: Relevance of Ventilatory Inefficiency
Brief Title: Comorbid Chronic Lung Disease on Heart Failure
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201701459B0
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Comorbid Chronic Lung Disease on Heart Failure
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure with chronic lung disease: Patients were recruited consecutively based on clinical assessment of risk factors for HF and echocardiographic evidence of systolic dysfunction or diastolic dysfunction. Risk factors for HF were defined as hypertension, atherosclerotic disease, obesity, chronic obstructive lung disease, metabolic syndrome, smoking, and family history of HF. In patients with normal LVEF (<50), diagnosis of diastolic dysfunction was based on echocardiographic parameters. Chronic lung disease (CLD) was defined as spirometry with obstructive lung disease or restrictive lung disease with accompanying clinical symptoms and signs included in the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
  Interventions: Diagnostic Test: cardiopulmonary exercise test
- Heart failure without chronic lung disease: Patients were recruited consecutively based on clinical assessment of risk factors for HF and echocardiographic evidence of systolic dysfunction or diastolic dysfunction. Risk factors for HF were defined as hypertension, atherosclerotic disease, obesity, chronic obstructive lung disease, metabolic syndrome, smoking, and family history of HF. In patients with normal LVEF (<50), diagnosis of diastolic dysfunction was based on echocardiographic parameters. Chronic lung disease (CLD) was defined as spirometry with obstructive lung disease or restrictive lung disease with accompanying clinical symptoms and signs included in the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria. HF patients who did not have chronic lung disease were assigned as a non-CLD group.
  Interventions: Diagnostic Test: cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: cardiopulmonary exercise test — Patients performed an upright graded bicycle exercise using a personalized protocol or performed a motorized treadmill exercise using a modified Bruce protocol. Peak VO2 and peak respiratory exchange ratio (RER) were defined as the highest 30-second average value obtained during exercise. The anaerobic threshold (AT) was determined by V-slope method. The VE(minute ventilation)/VCO2 (carbon dioxide production) at AT was calculated as the average VE/VCO2 for 1 minute during AT and immediately after AT. If AT could not be determined, the lowest VE/VCO2 was determined by averaging the three lowest consecutive 0.5-minute data points.

SUMMARY:
Comorbid chronic lung disease (CLD) increases mortality in heart failure (HF) patients. Understanding the predictors and pathophysiology of HF can improve the efficacy of HF treatment. This study evaluated the cardiopulmonary exercise test (CPET) results to identify significant predictors on long-term outcomes in HF patients with CLD.

DETAILED DESCRIPTION:
The CPET was administered in a cohort of 169 HF outpatients with exercise intolerance at a tertiary referral center between May 2007 and July 2010. A CLD was defined as abnormal spirometry accompanied by clinical symptoms and signs included in the Global Initiative for Chronic Obstructive Lung Disease criteria. The primary endpoint was defined as CV mortality or the first HF hospitalization. Totally 49 events occurred before the end of follow up in January 2018.

ELIGIBILITY:
Inclusion Criteria:

* outpatients ≥ 18 years of age, male or female.
* Patients with a diagnosis of heart failure with clinical symptoms and echocardiography evidence
* Patients received cardiopulmonary exercise test exams

Exclusion Criteria:

* Cannot tolerance exercise test due to muscular-skeletal disorder
* Cannot co-operate all functional studies
* Family reject to participate in this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 169 HF outpatients with exercise intolerance took the CPET at a tertiary referral center between May 2007 and July 2010. Patients were recruited consecutively based on clinical assessment of risk factors for HF and echocardiographic evidence of systolic dysfunction or diastolic dysfunction. In patients with normal LVEF (>=50), the diagnosis of diastolic dysfunction was based on echocardiographic parameters. Chronic lung disease (CLD) was defined as spirometry with obstructive lung disease or restrictive lung disease with accompanying clinical symptoms and signs included in the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria.
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants That Had Occurrence of the Composite Endpoint, Which is Defined as Either Cardiovascular (CV) Death or First Heart Failure (HF) Hospitalization | May, 2007 ~ January, 2018
  Number of participants that had occurrence of the composite endpoint, which is defined as either CV death or first HF hospitalization

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss with other investigators about individual participant data (IPD) sharing.